CLINICAL TRIAL: NCT00462202
Title: An Open Label Tolerability and Safety Study of KRX-101 (Sulodexide Gelcaps) for the Treatment of Type 2 Diabetic Nephropathic Patients With Persistent Microalbuminuria in Australia, New Zealand, and Hong Kong
Brief Title: Open Label Tolerability and Safety Study of KRX-101 in Australia, New Zealand, and Hong Kong
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Interim analysis of efficacy trial showed no drug efficacy.
Sponsor: Keryx Biopharmaceuticals (Industry)
Collaborators: Collaborative Study Group (CSG) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KRX 101-302
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Nephropathy
Keywords: Diabetes; Microalbuminuria; Proteinuria; Albuminuria; KRX-101; Sulodexide; Nephropathy; Keryx; Collaborative Study Group; Diabetic nephropathy with persistent microalbuminuria
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus; Proteinuria; Albuminuria; Kidney Diseases | interventions — glucuronyl glucosamine glycan sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sulodexide (Experimental): Open label extension to original trial
  Interventions: Drug: sulodexide

INTERVENTIONS:
Drug: sulodexide
  Other Names: KRX-101

SUMMARY:
The purpose of this study is to assess the tolerability and safety of KRX-101 in treating persistent microalbuminuria in type 2 diabetic patients who are also being treated with stable, maximum tolerated doses of either ACE inhibitors or A2 receptor blockers.

DETAILED DESCRIPTION:
Diabetes is one of the most common causes of end-stage renal disease (ESRD) in the U.S. and in many other developed nations. Despite advances in clinical care, including improvements in glycemic and blood pressure control, the number of new cases of diabetes-related ESRD continues to rise, especially in patients with type 2 diabetes.

The current standard of care for the prevention and treatment of diabetic renal disease includes screening all diabetic patients for microalbuminuria. Patients who test positive for microalbuminuria are then treated with either ACE inhibitors or A2 receptor blockers. Both of these classes of medication have been shown to reduce levels of microalbuminuria in some patient populations. This improvement in microalbuminuria has also shown a delay of progression to a number of other renal function problems, as well as a minimal delay in certain clinical events including ESRD.

Unfortunately, some patients achieve the majority of their therapeutic effect of ACE inhibitors or A2 receptor blockers within the first 6 months of therapy, and many of these patients continue to show persistent microalbuminuria. Therefore, these patients are at an increased risk of progressing to ESRD due to the lack of adequate benefit from their current medication.

Microalbuminuria has a straight-line relationship with adverse renal outcomes; therefore any level of reduction may have clinical benefit. It is reasonable to believe that patients who can reduce or have a complete remission of their microalbuminuria may also lessen the risk of progressing to ESRD. Thus, if KRX-101 is able to cause a reduction or complete remission of microalbuminuria to normoalbuminuria, patients may receive a significant clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and has successfully completed Keryx Study 101-301.
* Diagnosis of DM2 based on ADA criteria.
* Continued stable seated systolic blood pressure < 150 mmHg and diastolic blood pressure < 90 mmHg.
* Provide written informed consent to participate in the study.
* If female and of childbearing potential, must continue to be willing to use adequate contraception, as determined by the investigator, for the duration of the study.

Exclusion Criteria:

* Evidence of hepatic dysfunction including total bilirubin > 2.0 mg/dL (34 micromol/L) or liver enzymes > 3 times upper limit of normal.
* Unstable angina pectoris or New York Heart Association Class III or IV congestive heart failure.
* A history of any major medical condition, including but not limited to: aortic aneurysm; myocardial infarction, stroke, or other cardiovascular events in the past 3 months; gastrointestinal bleeding in the past 3 months; HIV; and other medical conditions deemed serious by the investigator. Active Hepatitis B or C (currently active disease defined as an abnormal liver biopsy or persistent, elevated transaminases, SGOT, SGPT).
* Any risk of bleeding, including a history of bleeding diathesis and a platelet count < 100,000/mm³.
* Active or metastatic cancer (note: superficial basal carcinoma of the skin is not an exclusion).
* Anticipated surgery within trial period.
* History of noncompliance to medical regimens in Keryx Study No.101-301.
* Participation in any experimental drug study in the past 60 days, except for KRX-101-301, prior to entry into the study, or plan to participate in any experimental drug study during the study period.
* Lactation, pregnancy, or an anticipated or planned pregnancy during the study period.
* Known allergy or intolerance to any heparin-like compounds.
* Patients with other specific renal diseases known to be the cause of nephropathy, and patients with other specific, clinically significant renal disease.
* Inability to give an informed consent or cooperate with the study personnel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Observed ACR level from the first visit to the end of study | 1 year
  Open label safety extension to assess long-term exposure to sulodexide (KRX-101) in patients with albumin and protein in their urine.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Atkins, MD, Study Director — Monash Medical Centre; Anne Reutens, MD, Principal Investigator — Monash Medical Center
Locations (1):
- Monash Medical Center, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No